CLINICAL TRIAL: NCT02415296
Title: Screening for Excessive Gambling Behaviors on the Internet (EDEIN Study). Study of the Database of French Online Gambling Sites.
Brief Title: Screening for Excessive Gambling Behaviors on the Internet
Acronym: EDEIN
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Université de Nantes (Other); ODJ (Observatoire des Jeux) (Unknown); ARJEL (Autorité de Régulation des Jeux En Ligne) (Other); MILDECA (Mission Interministérielle de Lutte contre les Drogues Et les Conduites Addictives) (Unknown); University of Paris 13 (Other); Institut de Recherche en Santé Publique, France (Other)
Responsible Party: Sponsor
Other Study IDs: PROG/10/124
Record Dates: First submitted 2015-04-01; First posted 2015-04-14 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Gambling, Pathological
Keywords: gambling disorder; screening model; online gambling; clinical validation
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- stage 1: French online gamblers.
  Interventions: Other: stage 1
- stage 2: Validation of problematic gamblers score on possible problematic gamblers.
  Interventions: Other: stage 2
- stage 3: 240 problematic gamblers.
  Interventions: Other: stage 3

INTERVENTIONS:
Other: stage 1 — The first stage of the project aims at providing a general description of the behaviour of French online gamblers, especially defining a typology of online gamblers.
  Groups: stage 1
Other: stage 2 — The second stage of the project aims at checking that the criteria selected in the first stage lead to a correct prediction whether the gambler is problematic or not. Particularly, this stage aims at determining the best possible score (calculated from gambling data) for defining the gambler's status.
  Groups: stage 2
Other: stage 3 — The third stage of the project aims at clinically validating the screening model. Result from the screening model will be compared to the diagnostic obtained with a clinical interview.
  Groups: stage 3

SUMMARY:
The Internet medium is particularly vector for gambling problems. Since the opening of the online gambling sector in France, no screening for excessive gambling behaviours is provided for by the law, although it is known that preventive actions are more effective if they are implemented early in the gambler's career.

The investigators propose to develop a model for screening excessive gambling practices based on the gambling behaviours observed on French gambling websites, coupled to a clinical validation. The objective is to lead to early preventive measures directed towards the more vulnerable gamblers and adapted for each type of gambling.

This study will therefore contribute to setting up an innovative measure of prevention, to inform and protect gamblers as early as possible.

ELIGIBILITY:
Inclusion Criteria:

* users of French online gambling websites
* users with active accounts
* users that have placed at least one bet during the last 12 months

Exclusion Criteria:

* minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be made up of users of French online gambling websites certified by the ARJEL within the context of law n° 2010-476 relative to opening the online gambling sector. Only active accounts, i.e. for which the gambler has placed at least one bet during the last 12 months, will be taken into account.
Sampling Method: Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2015-12-29 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Development of a model for screening excessive gambling practices based on the observation of the behaviour of online gamblers. | retrospective data collection over the past 12 months assessed at time 0

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital - IFAC, Nantes, France

REFERENCES:
- [Derived] Balem M, Perrot B, Hardouin JB, Thiabaud E, Saillard A, Grall-Bronnec M, Challet-Bouju G. Impact of wagering inducements on the gambling behaviors of on-line gamblers: A longitudinal study based on gambling tracking data. Addiction. 2022 Apr;117(4):1020-1034. doi: 10.1111/add.15665. Epub 2021 Sep 23. PMID 34374151
- [Derived] Perrot B, Hardouin JB, Costes JM, Caillon J, Grall-Bronnec M, Challet-Bouju G. Study protocol for a transversal study to develop a screening model for excessive gambling behaviours on a representative sample of users of French authorised gambling websites. BMJ Open. 2017 May 17;7(5):e014600. doi: 10.1136/bmjopen-2016-014600. PMID 28515192